CLINICAL TRIAL: NCT01635218
Title: Efficacy of Individualized Homeopathic Treatment for Moderate to Severe Depression in Peri- and Postmenopausal Women: a Randomized Placebo-controlled, Double-blind, Double-dummy, Study Protocol
Brief Title: Homeopathic Treatment for Depression in Peri- and Postmenopausal Women
Acronym: HOMDEP-MENOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Emma del Carmen Macías-Cortés, MD, PhD, MD, PhD, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HJM2030/12-A
Record Dates: First submitted 2012-06-30; First posted 2012-07-09 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-09

CONDITIONS: Moderate Depression; Menopausal and Postmenopausal Disorders
Keywords: Depression; Perimenopause; Postmenopause; Homeopathy
MeSH Terms: conditions — Depression | interventions — Materia Medica; Homeopathy; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individualized homeopathic treatment (Experimental): Selection of the individualized homeopathic remedy based on Hahnemann´s methodology after the case history of each patient.
  Interventions: Drug: Individualized homeopathic treatment
- Fluoxetine (Experimental): Selective serotonin reuptake inhibitor.
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Fluoxetine placebo plus individualized homeopathic placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Individualized homeopathic treatment — A single dose of the individualized homeopathic remedy in C-potency was dissolved in a 60 ml bottle of 30% alcohol-distilled water:15 drops PO two times per day following agitation plus fluoxetine-dummy loaded PO daily during 6 weeks. The homeopathic remedy could be changed at every follow-up (week 4) according to patient´s symptoms.
  Other Names: Homeopathic remedies; Homeopathic medicines
  Arms: Individualized homeopathic treatment
Drug: Fluoxetine — 20 mg per day PO during 6 weeks plus individualized homeopathic dummy-loaded (60 bottle of 30% alcohol-distilled water: 15 drops PO two times per day following agitation). The individualized homeopathic dummy-loaded was repeated at week 4.
  Other Names: Prozac
  Arms: Fluoxetine
Drug: Placebo — Fluoxetine placebo (capsules containing sucrose microgranules) PO daily during 6 weeks plus individualized homeopathic placebo (60 ml bottle of 30% alcohol-distilled water: 15 drops PO two times per day following agitation). The individualized homeopathic placebo was repeated at week 4.
  Other Names: Fluoxetine placebo; Individualized homeopathic placebo
  Arms: Placebo

SUMMARY:
The aim of this study was to determine whether individualized homeopathic treatment and fluoxetine are more efficient than placebo for moderate to severe depression in peri- and postmenopausal women.

DETAILED DESCRIPTION:
Perimenopausal period is characterized by an increased risk of depressive symptoms. Major depression is one of the most disabling medical conditions worldwide. At present, it is becoming more difficult to prove that antidepressants actually work better than placebo in clinical trials.Use of homeopathy to treat depression is widespread, but there is a lack of clinical trails about its efficacy in depression in peri- and postmenopausal women. Previous trials suggest that individualized homeopathic treatments improve depression in general population. The purpose of this study was to determine whether individualized homeopathic treatment and fluoxetine are more efficient than placebo for moderate depression in peri- and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Major depression according to DSM-IV
* Moderate to severe depression according to 17-item Hamilton Rating Scale for Depression (14-24 score)
* No current use of homeopathic treatment for depression or antidepressants or anxiolytic drugs 3 months prior to study entry
* Not be currently taking psychotherapy for at least 3 months before study entry
* Early transition to menopause defined by a change in cycle length of 7 days or longer in either direction from the participant´s own baseline for at least 2 cycles
* Late transition to menopause defined as 3 to 11 months of amenorrhea
* Postmenopausal stage defined by 12 months or more of amenorrhea
* Capability and willingness to give informed consent and to comply with the study procedures

Exclusion Criteria:

* Pregnancy or breastfeeding
* Other psychiatric disorders different from moderate to severe depression (severe depression, schizophrenia, psychotic disorders, bipolar affective disorders, suicide attempt)
* Alcohol or other substance abuse
* Known allergy to fluoxetine
* Cancer or hepatic diseases

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma del Carmen Macías-Cortés, MD, PhD, Principal Investigator — Hospital Juárez de México
Locations (1):
- Hospital Juárez de México, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Adler UC, Paiva NM, Cesar AT, Adler MS, Molina A, Padula AE, Calil HM. Homeopathic Individualized Q-Potencies versus Fluoxetine for Moderate to Severe Depression: Double-Blind, Randomized Non-Inferiority Trial. Evid Based Complement Alternat Med. 2011;2011:520182. doi: 10.1093/ecam/nep114. Epub 2011 Jun 8. PMID 19687192
- [Background] Frank E, Prien RF, Jarrett RB, Keller MB, Kupfer DJ, Lavori PW, Rush AJ, Weissman MM. Conceptualization and rationale for consensus definitions of terms in major depressive disorder. Remission, recovery, relapse, and recurrence. Arch Gen Psychiatry. 1991 Sep;48(9):851-5. doi: 10.1001/archpsyc.1991.01810330075011. PMID 1929776
- [Background] Hale GE, Zhao X, Hughes CL, Burger HG, Robertson DM, Fraser IS. Endocrine features of menstrual cycles in middle and late reproductive age and the menopausal transition classified according to the Staging of Reproductive Aging Workshop (STRAW) staging system. J Clin Endocrinol Metab. 2007 Aug;92(8):3060-7. doi: 10.1210/jc.2007-0066. Epub 2007 Jun 5. PMID 17550960
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Murray CJ, Lopez AD. Evidence-based health policy--lessons from the Global Burden of Disease Study. Science. 1996 Nov 1;274(5288):740-3. doi: 10.1126/science.274.5288.740. No abstract available. PMID 8966556
- [Background] Greenberg PE, Stiglin LE, Finkelstein SN, Berndt ER. The economic burden of depression in 1990. J Clin Psychiatry. 1993 Nov;54(11):405-18. PMID 8270583
- [Background] Williams LM, Rush AJ, Koslow SH, Wisniewski SR, Cooper NJ, Nemeroff CB, Schatzberg AF, Gordon E. International Study to Predict Optimized Treatment for Depression (iSPOT-D), a randomized clinical trial: rationale and protocol. Trials. 2011 Jan 5;12:4. doi: 10.1186/1745-6215-12-4. PMID 21208417
- [Background] Simon GE, VonKorff M, Barlow W. Health care costs of primary care patients with recognized depression. Arch Gen Psychiatry. 1995 Oct;52(10):850-6. doi: 10.1001/archpsyc.1995.03950220060012. PMID 7575105
- [Background] Cohen LS, Soares CN, Vitonis AF, Otto MW, Harlow BL. Risk for new onset of depression during the menopausal transition: the Harvard study of moods and cycles. Arch Gen Psychiatry. 2006 Apr;63(4):385-90. doi: 10.1001/archpsyc.63.4.385. PMID 16585467
- [Background] Freeman EW, Sammel MD, Lin H, Nelson DB. Associations of hormones and menopausal status with depressed mood in women with no history of depression. Arch Gen Psychiatry. 2006 Apr;63(4):375-82. doi: 10.1001/archpsyc.63.4.375. PMID 16585466
- [Background] Freeman EW, Sammel MD, Liu L, Gracia CR, Nelson DB, Hollander L. Hormones and menopausal status as predictors of depression in women in transition to menopause. Arch Gen Psychiatry. 2004 Jan;61(1):62-70. doi: 10.1001/archpsyc.61.1.62. PMID 14706945
- [Background] Rapkin AJ. Vasomotor symptoms in menopause: physiologic condition and central nervous system approaches to treatment. Am J Obstet Gynecol. 2007 Feb;196(2):97-106. doi: 10.1016/j.ajog.2006.05.056. PMID 17306645
- [Background] Fava M, Davidson KG. Definition and epidemiology of treatment-resistant depression. Psychiatr Clin North Am. 1996 Jun;19(2):179-200. doi: 10.1016/s0193-953x(05)70283-5. PMID 8827185
- [Background] Davidson JR, Crawford C, Ives JA, Jonas WB. Homeopathic treatments in psychiatry: a systematic review of randomized placebo-controlled studies. J Clin Psychiatry. 2011 Jun;72(6):795-805. doi: 10.4088/JCP.10r06580. PMID 21733480
- [Background] Adler UC, Kruger S, Teut M, Ludtke R, Bartsch I, Schutzler L, Melcher F, Willich SN, Linde K, Witt CM. Homeopathy for depression--DEP-HOM: study protocol for a randomized, partially double-blind, placebo controlled, four armed study. Trials. 2011 Feb 14;12:43. doi: 10.1186/1745-6215-12-43. PMID 21320338
- [Background] Freeman MP, Mischoulon D, Tedeschini E, Goodness T, Cohen LS, Fava M, Papakostas GI. Complementary and alternative medicine for major depressive disorder: a meta-analysis of patient characteristics, placebo-response rates, and treatment outcomes relative to standard antidepressants. J Clin Psychiatry. 2010 Jun;71(6):682-8. doi: 10.4088/JCP.10r05976blu. PMID 20573327
- [Background] Linde K, Melchart D. Randomized controlled trials of individualized homeopathy: a state-of-the-art review. J Altern Complement Med. 1998 Winter;4(4):371-88. doi: 10.1089/acm.1998.4.371. PMID 9884175
- [Background] Thompson TD, Weiss M. Homeopathy--what are the active ingredients? An exploratory study using the UK Medical Research Council's framework for the evaluation of complex interventions. BMC Complement Altern Med. 2006 Nov 13;6:37. doi: 10.1186/1472-6882-6-37. PMID 17101037
- [Background] Dean ME, Coulter MK, Fisher P, Jobst K, Walach H; Delphi Panel of the CONSORT Group. Reporting data on homeopathic treatments (RedHot): a supplement to CONSORT*. Forsch Komplementmed. 2006 Dec;13(6):368-71. doi: 10.1159/000097073. Epub 2006 Dec 21. PMID 17200612
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomized trials. Open Med. 2010;4(1):e60-8. Epub 2010 Mar 24. No abstract available. PMID 21686296
- [Background] Ludtke R, Rutten ALB. The conclusions on the effectiveness of homeopathy highly depend on the set of analyzed trials. J Clin Epidemiol. 2008 Dec;61(12):1197-1204. doi: 10.1016/j.jclinepi.2008.06.015. Epub 2008 Oct 1. PMID 18834714
- [Background] Bordet MF, Colas A, Marijnen P, Masson J, Trichard M. Treating hot flushes in menopausal women with homeopathic treatment--results of an observational study. Homeopathy. 2008 Jan;97(1):10-5. doi: 10.1016/j.homp.2007.11.005. PMID 18194760
- [Background] Shang A, Huwiler-Muntener K, Nartey L, Juni P, Dorig S, Sterne JA, Pewsner D, Egger M. Are the clinical effects of homoeopathy placebo effects? Comparative study of placebo-controlled trials of homoeopathy and allopathy. Lancet. 2005 Aug 27-Sep 2;366(9487):726-32. doi: 10.1016/S0140-6736(05)67177-2. PMID 16125589
- [Background] Mulrow CD, Williams JW Jr, Chiquette E, Aguilar C, Hitchcock-Noel P, Lee S, Cornell J, Stamm K. Efficacy of newer medications for treating depression in primary care patients. Am J Med. 2000 Jan;108(1):54-64. doi: 10.1016/s0002-9343(99)00316-2. PMID 11059441
- [Background] Dawson MY, Michalak EE, Waraich P, Anderson JE, Lam RW. Is remission of depressive symptoms in primary care a realistic goal? A meta-analysis. BMC Fam Pract. 2004 Sep 7;5:19. doi: 10.1186/1471-2296-5-19. PMID 15353006
- [Derived] Macias-Cortes EDC, Llanes-Gonzalez L, Aguilar-Faisal L, Asbun-Bojalil J. Response to Individualized Homeopathic Treatment for Depression in Climacteric Women with History of Domestic Violence, Marital Dissatisfaction or Sexual Abuse: Results from the HOMDEP-MENOP Study. Homeopathy. 2018 Aug;107(3):202-208. doi: 10.1055/s-0038-1654709. Epub 2018 Jun 5. PMID 29871025
- [Derived] Macias-Cortes ED, Llanes-Gonzalez L, Aguilar-Faisal L, Asbun-Bojalil J. Is metabolic dysregulation associated with antidepressant response in depressed women in climacteric treated with individualized homeopathic medicines or fluoxetine? The HOMDEP-MENOP Study. Homeopathy. 2017 Feb;106(1):3-10. doi: 10.1016/j.homp.2016.11.002. Epub 2017 Jan 10. PMID 28325221
- [Derived] Macias-Cortes Edel C, Llanes-Gonzalez L, Aguilar-Faisal L, Asbun-Bojalil J. Individualized homeopathic treatment and fluoxetine for moderate to severe depression in peri- and postmenopausal women (HOMDEP-MENOP study): a randomized, double-dummy, double-blind, placebo-controlled trial. PLoS One. 2015 Mar 13;10(3):e0118440. doi: 10.1371/journal.pone.0118440. eCollection 2015. PMID 25768800 (Retraction: PMID 32324840 PLoS One. 2020 Apr 23;15(4):e0232415)
- [Derived] Macias-Cortes Edel C, Aguilar-Faisal L, Asbun-Bojalil J. Efficacy of individualized homeopathic treatment and fluoxetine for moderate to severe depression in peri- and postmenopausal women (HOMDEP-MENOP): study protocol for a randomized, double-dummy, double-blind, placebo-controlled trial. Trials. 2013 Apr 23;14:105. doi: 10.1186/1745-6215-14-105. PMID 23782520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a public, academic and research hospital in Mexico City. Participants were recruited since March 2012 until December 2013. The recruitment methods included advertisements through internet, community groups,liaisons with health professionals, posters and brochures distributed among hospital population.
Pre-assignment Details: Five hundred thirty-four women seeking medical care for menopausal complaints were interviewed and screened. Four hundred and one women did not meet inclusion criteria and were excluded: no depression (44), mild depression (150), severe depression and/or attempt of suicide (43), did not meet other inclusion criteria (164).
Period: Overall Study
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Started | 44 | 46 | 43
Completed | 41 | 39 | 37
Not Completed | 3 | 7 | 6
Not completed — Lost to Follow-up | 3 | 7 | 6

BASELINE CHARACTERISTICS:
Population: All patientes under randomization were included in the primary efficacy population (intention-to-treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 43 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (6.4) | 49.2 (5.3) | 48.8 (5.8) | 49 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 43 | 133
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 46 | 43 | 133
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 44 | 46 | 43 | 133
Baseline score in 17-item Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: Units in Hamilton Scale] — A total score in 17-item Hamilton Scale for Depression was assessed for this study. It ranges from 0 (no depression) up to 52 (most severe depression). A score < or = 7 is considered normal, 7 - 13 (mild depression), 14 - 24 (moderate to severe depression), > 24 (severe depression). The score of the 17 items was summed.
  The score presented here is the baseline score of Hamilton Scale, the final score after the 6 weeks treatment is presented in Outcomes measure data table.
  Units in Hamilton Scale | 21.2 (2.7) | 20.6 (2.9) | 20.7 (3.1) | 20.8 (2.9)
Baseline score in Beck Depression Inventory [Mean (Standard Deviation); unit: Units in Beck Depression Inventory] — Beck Depression Inventory is a 21-question multiple-choice self-report inventory. For this study a total score range was assessed: 0 (without depression) up to 63 (most severe depression): 0 - 8 is considered normal, 9 - 18 (mild to moderate depression), 19 - 28 (moderate to severe depression), > 29 (severe depression). The score of the 21 questions was summed.
  The score presented here is the baseline score of BDI, the final score after the 6 weeks treatment is presented in the Outcome measure data table.
  Units in Beck Depression Inventory | 26.3 (7.2) | 25.0 (7.8) | 27.0 (9.0) | 26.1 (8.0)
Baseline score in Greene Climacteric Scale [Mean (Standard Deviation); unit: Units in Greene Climacteric Scale] — Greene Climacteric Scale is intended to be a standard measure of core climacteric symptoms. For this study a total range was assessed: 0 (without climacteric symptoms) up to 63 (most severe climacteric symptoms). The scale measures four separate sub-scales (anxiety, depression, somatic symptoms and sexual function). The score of the four sub-scales was summed. A total score of 0 -10 is considered without symptoms, 11 - 29 (mild symptoms), 30 - 49 (moderate symptoms) and > 50 (severe symptoms).
  The score presented here is the baseline score of Greene Climacteric Scale before treatment.
  Units in Greene Climacteric Scale | 35.3 (8.5) | 33.5 (10.1) | 37.9 (11.5) | 35.5 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 17-item Hamilton Rating Scale for Depression at 6 Weeks.
Description: 17-item Hamilton Rating Scale for Depression (HRSD) is a well-known standardized scale used worldwide to assess severity of depression. Score ranges from 0 (no depression) up to 52 (maximum depression severity). A total score in HRSD was assessed at baseline and after six weeks of treatment. For this study the change was calculated as the later time point (total score in 17- HRSD at 6 weeks) minus the earlier time point (total score at baseline). A score < or = 7 is considered normal, 7 - 13 (mild depression), 14 - 24 (moderate to severe depression), > 24 (severe depression).
Time Frame: Baseline and 6 weeks
Population: All patients under randomization were included in the primary efficacy population (intention-to-treat population), regardless whether or not they adhered to the treatment protocol or provided complete data sets.The mean and SD presented in outcome measure data table are the final scores in Hamilton Scale after 6 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Units in Hamilton Scale
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Number analyzed (Participants) | 44 | 46 | 43
Units in Hamilton Scale | 9.9 (3) | 11.7 (3.7) | 15 (3.7)
Statistical Analysis 1: Comparison: Individualized Homeopathic Treatment vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA — The ANOVA result (p<0.05)suggests rejecting the global null hypothesis.Bonferroni post-hoc test was used to determine which means differ among groups; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [3.1 to 7.0], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [1.31 to 5.25], Standard Error of Mean 0.81

2. Secondary Outcome: Change From Baseline in Beck Depression Inventory at 6 Weeks.
Description: Beck Depression Inventory (BDI) is a 21-question multiple-choice self-report inventory that assess severity of depression. A total score range was assessed at baseline and after six weeks of treatment. A score 0 (without depression) up to 63 (most severe depression). For this study the change was calculated as the later time point (total score in BDI at 6 weeks) minus the earlier time point (total score in BDI at baseline). A score 0 - 8 is considered normal, 9 - 18 (mild to moderate depression), 19 - 28 (moderate to severe depression), > 29 (severe depression).
Time Frame: Baseline and 6 weeks
Population: All patients under randomization were included in the primary efficacy population (intention-to-treat population) regardless whether or not they adhered to the treatment protocol or provided complete data sets. The mean and SD presented here in the Outcome measure data table are the final scores after 6 weeks treatment.
Measure: Mean (Standard Deviation); unit: Units in Beck Depression Inventory
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Number analyzed (Participants) | 44 | 46 | 43
Units in Beck Depression Inventory | 12 (6.1) | 14.2 (7.8) | 15.5 (8.8)
Statistical Analysis 1: Comparison: Individualized Homeopathic Treatment vs Placebo; Test type: Superiority or Other; p = 0.14, ANOVA — The statistical significant ANOVA result (p<0.05) suggests rejecting the global null hypothesis.Bonferroni post-hoc test was used to determine which means differ among groups; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-0.73 to 7.61], Standard Error of Mean 1.71
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority or Other; p = 0.99, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [-2.93 to 5.5], Standard Error of Mean 1.73

3. Secondary Outcome: Responder Rates at 6 Weeks.
Description: 17-item Hamilton Rating Scale for Depression is a well-known standardized scale used worldwide to assess severity of depression. Score ranges from 0 (no depression) up to 52 (maximum depression severity). A total score in 17-item Hamilton Scale for Depression was assessed for this study. It ranges from 0 (no depression) up to 52 (most severe depression). A score < or = 7 is considered normal, 7 - 13 (mild depression), 14 - 24 (moderate to severe depression), > 24 (severe depression). Responder rate definition: a decrease of 50% or more from baseline score using 17-item Hamilton Rating Scale for Depression after six weeks treatment.
Time Frame: 6 weeks
Population: All patients under randomization were included in the primary efficacy population (intention-to-treat population) regardless whether or not they adhered to the treatment protocol or provided complete data sets.
Measure: Number; unit: participants with a decrease >50% in HS
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Number analyzed (Participants) | 44 | 46 | 43
participants with a decrease >50% in HS | 24 | 19 | 5
Statistical Analysis 1: Comparison: Individualized Homeopathic Treatment vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.03 to 0.34]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 0.19, 95% CI 2-sided [0.06 to 0.56]

4. Secondary Outcome: Change From Baseline in Greene´s Scale at 6 Weeks.
Description: Greene Climacteric Scale (GS) is intended to be a standard measure of core climacteric symptoms. For this study a total range was assessed at baseline and after six weeks of treatment. A total score 0 (without climacteric symptoms) up to 63 (most severe climacteric symptoms). The change was calculated as the later time point (total score in GS at 6 weeks) minus the earlier time point (total score at baseline).The scale measures four separate sub-scales (anxiety, depression, somatic symptoms and sexual function). The score of the four sub-scales was summed. A total score of 0 -10 is considered without symptoms, 11 - 29 (mild symptoms), 30 - 49 (moderate symptoms) and > 50 (severe symptoms).
Time Frame: Baseline and 6 weeks
Population: All patients under randomization were included in the primary efficacy population (intention-to-treat population) regardless whether or not they adhered to the treatment protocol or provided complete data sets.The mean and SD presented here in the Outcome measure data table are the final scores after 6 weeks treatment.
Measure: Mean (Standard Deviation); unit: Units in Green Scale
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Number analyzed (Participants) | 44 | 46 | 43
Units in Green Scale | 18.1 (7.8) | 23.1 (12.3) | 26.8 (11.7)
Statistical Analysis 1: Comparison: Individualized Homeopathic Treatment vs Placebo; Test type: Superiority or Other; p = 0.002, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [2.72 to 14.52], Standard Error of Mean 2.42
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority or Other; p = 0.424, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-2.33 to 9.6], Standard Error of Mean 2.37

5. Secondary Outcome: Remission Rates at 6 Weeks
Description: 17-item Hamilton Rating Scale for Depression is a well-known standardized scale used worldwide to assess severity of depression. Score ranges from 0 (no depression) up to 52 (maximum depression severity). A total score in 17-item Hamilton Scale for Depression was assessed for this study. It ranges from 0 (no depression) up to 52 (most severe depression). A score < or = 7 is considered normal, 7 - 13 (mild depression), 14 - 24 (moderate to severe depression), > 24 (severe depression). Remission rate definition: 17-item Hamilton Rating Scale for Depression score < 7 points after 6 weeks of treatment.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Number; unit: participants with a score of < 7 in HS
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Number analyzed (Participants) | 44 | 46 | 43
participants with a score of < 7 in HS | 7 | 7 | 2
Statistical Analysis 1: Comparison: Individualized Homeopathic Treatment vs Placebo; Test type: Superiority or Other; p = 0.10, Chi-squared; Odds Ratio (OR) = 0.26, 95% CI [0.05 to 1.32]
Statistical Analysis 2: Comparison: Fluoxetine vs Placebo; Test type: Superiority or Other; p = 0.11, Chi-squared; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.05 to 1.39]

ADVERSE EVENTS:
Time Frame: During study duration and 2 weeks after the final dose (8 weeks).
Description: Daily patient's questionnaire and medical examination at each follow-up.
Groups:
- Fluoxetine: Selective serotonin reuptake inhibitor.
  Fluoxetine: 20 mg per day PO during 6 weeks plus individualized homeopathic dummy-loaded (60 bottle of 30% alcohol-distilled water: 15 drops PO two times per day following agitation). The individualized homeopathic dummy-loaded could be repeated at week 4.
Arm/Group | Individualized Homeopathic Treatment | Fluoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 0/43
Other Adverse Events (participants affected / at risk) | 19/44 | 24/46 | 16/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Homeopathic Treatment (N=44) | Fluoxetine (N=46) | Placebo (N=43)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 6 (6) | 5 (5)
Insomnia (Psychiatric disorders) | 6 (6) | 5 (5) | 6 (6)
Anxiety (Psychiatric disorders) | 4 (4) | 8 (8) | 2 (2)
Dizziness (General disorders) | 4 (4) | 5 (5) | 4 (4)
Fatigue (General disorders) | 5 (5) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No